CLINICAL TRIAL: NCT03289637
Title: Supplementation With Vitamin D to Patients With Heart Failure. Effects on Symptoms, Quality-of-life and Disease Processes.
Brief Title: Supplementation With Vitamin D to Patients With Heart Failure (D-Heart).
Acronym: D-Heart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Urban Alehagen, Professor, MD., Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-88538-Sw
Record Dates: First submitted 2017-09-06; First posted 2017-09-21 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Double blind, parallel, placebo controlled study
Who Masked: Participant, Care Provider
Masking Description: Neither the participant, nor the care provider will be informed if active supplementation or placebo will be given, nor will blood sample results be open for care provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): In the group randomised to active treatment and with a screening level of 25-OH-vitamin D 25-50nmol/L an intervention with 1600IE daily of vitamin D will be given.
  In those randomised to active treatment and with a screening level of 25-OH-vitamin D of <25nmol/L, an intervention of 2400IE of vitamin D will be given.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): In the group randomised to placebo and with a screening level of 25-OH-vitamin D <50 mol/L, the participants will be given placebo.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D intervention tested against placebo in a population with heart failure and a 25-OH-vitamin D level<50nmol/L at screening

SUMMARY:
In 200 patients with documented systolic heart failure give supplementation with vitamin D in those with a 25-OH- vitamin D < 50nmol/L - or placebo.

In those with a vitamin D level <25nmol/L a substitution of 2400IU will be given, and in those with a vitamin D level 25-50nmol/L a substitution of 1600IU will be given.

Intervention time 12 months. Biomarkers of heart function, quality of life, and hospitalisation will be analysed.

DETAILED DESCRIPTION:
In a population with a systolic heart failure with an EF<40%, the levels of vitamin D will be analysed. In those with a 25-OH-vitamin D level <50nmol/L the patients that accept participation, will be randomised into active supplementation as described below, or placebo.

* In those with a 25-OH-vitamin D level <25nmol/L there will be a supplementation of 2400IU daily
* In those with a vitamin D level 25-50nmol/L there will be a supplementation of 1600IU daily,
* or placebo. Thus based on the basal level of vitamin D the screened patients will either be excluded due to high level of vitamin D, or given one ot the two options of vitamin D dosage based on the basal patient level - or placebo.

The intervention time will be 12 months. In the project 200 heart failure patients will be included. Blood samples including heart failure biomarkers, and biomarkers for inflammation and oxidative stress will be drawn at 3,6, 9 and 12 months.

Health related quality of life will be evaluated by use of Euro-QoL-5D Minnesota Living with Heart Failure.Patient Health Questionnaire-9 Multidimensional Fatigue Inventory 20 questionnaire, as also hospitalisation during the project time.

Cardiac function according to echocardiography will be analysed at start, and study end.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented and stable systolic heart failure and connected to an outpatient clinic at the Dept of Cardiology in Linköping, or Jönköping, Sweden, and with a 25-OH-vitamin D <50nmol/L

Exclusion Criteria:

* Patients with unstable heart failure
* Patients with significant valvular disease, or ischemic heart disease planned for operation
* Patients with significant renal or /and liver impairment.
* Patients that do not understand that study information, or that are not willing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the composite endpoint for heart failure | Follow-up 12 months after stop of intervention
  Reduction in biomarkers for heart failure(Nt-proBNP, Copeptin, MR-proADM and Chromogranin A) and in hospitalisation that comprised the composite endpoint

SECONDARY OUTCOMES:
Influence on quality of life in patients with heart failure by the intervention | Follow-up 12 months after stop of intervention
  Effect on health related quality of life as measured by the Euro-QoL-5D Minnesota Living with Heart Failure. Patient Health Questionnaire-9 Multidimensional Fatigue Inventory 20 questionnaires

OTHER OUTCOMES:
Influence on quality of life in patients with heart failure by the intervention | Follow-up 12 months after termination of the intervention
  Effect on health related quality of life as measured by Minnesota Living with Heart Failure
Influence on symptoms of depression in patients with heart failure by the intervention | Follow-up 12 months after termination of intervention
  Patient Health Questionnaire-9 (PHQ-9)
Influence on perceived fatigue in patients with heart failure by the intervention | Follow-up 12 months after termination of the intervention
  Effect on as measured using the Multidimensional Fatigue Inventory 20

CONTACTS AND LOCATIONS:
Overall Officials: Urban Alehagen, Prof, Principal Investigator — University of Linköping
Locations (1):
- Dept of Cardiology, University Hospital of Linköping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No